CLINICAL TRIAL: NCT01140126
Title: A Phase I, Open-label, Single-dose, Dose-escalation Study to Evaluate the Safety and Pharmacokinetics of the UB-421 Antibody in Asymptomatic HIV-1 Infected Adults
Brief Title: Study to Evaluate Safety and Pharmacokinetics of UB-421 Antibody in HIV-1 Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Biomedical (Industry)
Responsible Party: Wing Wai Wong, M.D., Taipei Veterans General Hospital (TVGH), Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBI Protocol A101; Protocol A101-HIV (Other: UBI-Asia)
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: HIV-1 Infection in Adults (Asymptomatic)
Keywords: HIV-1, CD4, antibody, immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antibody (UB-421) (Experimental)
  Interventions: Drug: Antibody UB-421

INTERVENTIONS:
Drug: Antibody UB-421 — Single intravenous infusion at day 0 of a liquid dose of 1, 5, 10 or 25 mg/kg body weight.

SUMMARY:
The purpose of this Phase I study is to determine whether the antibody (UB-421), targeting the HIV-1 receptor on the CD4 molecule (domain 1) of T-lymphocytes and monocytes, is safe and well tolerated when administered to asymptomatic HIV-1 infected adults by intravenous infusion and to assess pharmacokinetic parameters of the antibody in blood and on cells. The neutralizing activity of UB-421 blocks HIV-1 from binding to its receptor on CD4-positive cells; thus, UB-421 functions as an immunotherapeutic intervention to prevent HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic, treatment-naive, HIV-1 seropositive
* CD4+ T cell count >350 cells/cubic millimeter
* HIV-1 viral load >5,000 copies/mL
* Other inclusion criteria apply

Exclusion Criteria:

* Active infection requiring immediate therapy (except HIV-1)
* Prior participation in any HIV vaccine trial
* Previous exposure to a monoclonal antibody
* Use of immunomodulating drugs or systemic chemotherapy
* Other exclusion criteria apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of a single intravenous infusion at escalating doses of UB-421. | Screen, treatment & follow-up: 62 to 90 days

SECONDARY OUTCOMES:
To determine pharmacokinetic parameters of a single intravenous infusion at escalating doses of UB-421. | Screen, treatment & follow-up: 62 to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Wing Wai Wong, M.D., Principal Investigator — Taipei Veterans General Hospital (TVGH), Taiwan; Hung Chin Tsai, M.D., Principal Investigator — Kaohsiung Veterans General Hospital (KVGH), Taiwan
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital (TVGH), Taipei, Beitou District
  - Kaohsiung Veterans General Hospital (KVGH), Kaohsiung City, Zuoying District

REFERENCES:
- [Background] Wang CY, Sawyer LS, Murthy KK, Fang X, Walfield AM, Ye J, Wang JJ, Chen PD, Li ML, Salas MT, Shen M, Gauduin MC, Boyle RW, Koup RA, Montefiori DC, Mascola JR, Koff WC, Hanson CV. Postexposure immunoprophylaxis of primary isolates by an antibody to HIV receptor complex. Proc Natl Acad Sci U S A. 1999 Aug 31;96(18):10367-72. doi: 10.1073/pnas.96.18.10367. PMID 10468614